CLINICAL TRIAL: NCT01730508
Title: A MULTICENTER, PROSPECTIVE, OBSERVATIONAL, NON-INTERVENTIONAL COHORT STUDY IN CHINESE SUBJECTS WITH HBeAg NEGATIVE CHRONIC HEPATITIS B (CHB) RECEIVING THERAPY WITH PEGINTERFERON ALFA
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) in Chinese Patients With HBeAg Negative Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28516
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Hepatitis B Participants: Hepatitis B e antigen (HBeAg) chronic hepatitis B (CHB) participants who received treatment with pegylated interferon alfa (peginterferon alfa) according to China labeling and China standard of care and were followed up to 1 year after treatment cessation.
  Interventions: Drug: Pegylated Interferon Alfa (Peginterferon Alfa)

INTERVENTIONS:
Drug: Pegylated Interferon Alfa (Peginterferon Alfa) — Peginterferon alfa dosing and treatment duration are at the discretion of the investigator in accordance with China clinical practice and local labeling.
  Other Names: Pegasys

SUMMARY:
This multicenter, prospective, observational study will evaluate the use in clinical practice and the efficacy and safety of Pegasys (peginterferon alfa-2a) in Chinese participants with HBeAg negative chronic hepatitis B. Participants receiving Pegasys according to the local label will be followed for the duration of their treatment and for one year after cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Treatment with Pegasys according to label and standard clinical practice
* HBeAg negative serologically proven chronic hepatitis B with or without cirrhosis
* Serum alanine aminotransferase (ALT) > upper limit of normal (ULN) but </= 10 x ULN
* Hepatitis B Virus (HBV) DNA >/= 2000 IU/mL

Exclusion Criteria:

* Contraindications to Pegasys as detailed in the label
* Co-infection with hepatitis A, hepatitis C or HIV
* Pregnant or lactating women
* Participants should not receive concomitant therapy with telbivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants with HBeAg negative chronic hepatitis B receiving treatment with Pegasys
Sampling Method: Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of sustained suppression of HBV DNA <2000 IU/mL one year after treatment cessation | approximately 4 years

SECONDARY OUTCOMES:
Incidence of suppression of HBV DNA <2000 IU/mL at the end of treatment and 6 months post-treatment | approximately 4 years
Incidence of HBV DNA undetectable (<400 IU/mL) at the end of treatment and 1 year post-treatment | approximately 4 years
Incidence of HBsAg loss/seroconversion | approximately 4 years
Incidence of normalization of serum ALT levels | approximately 4 years
Dosage/schedule of Pegasys treatment in real-life clinical setting | approximately 4 years
Clinical/demographic patient characteristics at initiation of treatment | approximately 4 years
Safety: Incidence of adverse events | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (88):
- China (88):
  - The Fifth Hospital of Shijiazhuang, Baoding
  - Beijing Ditan Hospital, Beijing
  - Beijing 302 Hospital; No. 2 Infectious Disease Section, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing You An Hospital; Digestive Dept, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Hepatobiliary Hospital, Changchun
  - Peoples Hospital of Hunan Province, Changsha
  - The Third Xiangya Hospital Of Central South University, Changsha
  - Changzhou 3rd People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital, Chongqing Medical University, Chongqing
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Southwest Hospital , Third Military Medical University, Chongqing
  - 6th Hospital of Dalian City, Dalian
  - The First People's Hospital of Foshan, Foshan
  - The First People's Hospital of Shunde, Foushan
  - Fuzhou Infectious Diseases Hospital, Fuzhou
  - The Eighth People's Hospital of Guangzhou, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - Guangdong Provincial Traditional Chinese Medicine Hospital, Guangzhou
  - Hainan provincial people's hospital, Haikou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University(First Hospital of Zhejiang, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - 211 Military Hospital of China, Harbin
  - The 4th Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huai'an No 4 People's Hospital, Huai'an
  - Jiangmen Wuyi Traditional Chinese Medicine Hospital, Jiangmen
  - Jiangyin People's Hospital, Jiangyin
  - Jinan Infectious Diseases Hospital, Jinan
  - Third people's Hospital of Kunming City, Kunming
  - The Second Gansu Province General Hospital, Lanzhou
  - The First People's Hospital of Lian Yun Gang, Lianyungang
  - Liuzhou Hospital of Traditional Chinese Medicine, Liuchow
  - Affiliated Hospital of Luzhou medical college, Luzhou
  - The Ninth Hospital of Nanchang, Nanchang
  - Nanjing No.2 Hospital; Liver Disease Department, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The 81st Hospital of P.L.A., Nanjing
  - Ruikang Hospital Affiliated to Guangxi University of Chinese Medicine, Nanning
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Ningbo No.2 Hospital, Ningbo
  - Ordos No.2 Hospital, Ordos
  - QingDao Infection Diseases Hospital, Qingdao
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - No.3 people's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - Shanghai Huangpu District Central Hospital, Shanghai
  - The First Affiliated Hospital, Shantou University, Shantou
  - Shengjing Hospital of China Medical University, Shenyang
  - Shenyang Sixth People's Hospital （Shenyang Infectious Disease Hospital）, Shenyang
  - Shenzhen Donghu Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Bethune International Peace Hospital of PLA, Shijiazhuang
  - Suining Central Hospital, Suining
  - The Fifth People's Hospital Suzhou; Infectious Disease, Suzhou
  - The Third Hospital of Taiyuan (Taiyuan Infectious Diseases Hospital), Taiyuan
  - Jiangsu Taizhou People's Hospital, Taizhou
  - Tianjin Infectious Disease Hospital, Tianjin
  - Dagang Oil Field General Hospital, Tianjin
  - Xinjiang Uygur Autonomous Region Hospital of Chinese Traditional Medicine, Ürümqi
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - Wenzhou Hospital of Traditional Chinese Medicine, Wenzhou
  - Ruian People's Hospital, Wenzhou
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - Wuxi No.5 People's Hospital, Wuxi
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - Xiamen Hospital of T.C.M, Xiamen
  - Xingtai People's Hospital, Xingtai
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Yancheng City No.1 People's Hospital, Yancheng
  - Yangzhou Third People's Hospital, Yangzhou
  - Central People's Hospital of Yichang, Yichang
  - Chinese medicine hospital of Zhaoqing City, Zhaoqing
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhenjiang Third People's Hospital, Zhenjiang
  - Zhoushan Hospital, Zhoushan
  - Zhuhai People's Hospital, Zhuhai

REFERENCES:
- [Derived] Chen X, Mao Q, Xie Y, Dou X, Xie Q, Sheng J, Gao Z, Zhou X, Liu Y, Zheng H, Zhang S, Li S, Zhu F, Xu Y, Zhang M, Hu Y, Chen X, Huang Y, Ren H, Jia J. A Potential Functional Cure in Chinese HBeAg-negative Chronic Hepatitis B Patients Treated with Peg-interferon Alpha-2a. J Clin Transl Hepatol. 2019 Sep 28;7(3):249-257. doi: 10.14218/JCTH.2019.00016. Epub 2019 Aug 20. PMID 31608217